CLINICAL TRIAL: NCT06322121
Title: Clarifying the Vascular Aspects of Dementia; Natural History Study
Brief Title: Vascular Aspects in Dementia: Part 2
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, svanrooden, dr. Principal Investigator, Leiden University Medical Center
Other Study IDs: NL83653.058.23
Record Dates: First submitted 2023-12-11; First posted 2024-03-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 ml saliva for APOE genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Dementia patients: Patients with a dementia diagnosis; probable Alzheimer or mixed-type dementia
  Interventions: Other: MRI
- MCI patients: Patients with a MCI diagnosis; patients demonstrating cognitive deficits on neuropsychological testing but not fulfilling the criteria for dementia.
  Interventions: Other: MRI
- SCI patients: Patients not demonstrating cognitive deficits on neuropsychological testing are classified as SCI
  Interventions: Other: MRI
- Controls: Control subject without cognitive complaints
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Assessment of vascular reactivity and CAA/SVD MRI markers

SUMMARY:
Cerebral amyloid angiopathy (CAA), a common cerebrovascular small vessel disease (SVD), is a frequently (98%) found co-morbidity at autopsy in patients with Alzheimer's disease (AD). Current in vivo hallmarks of CAA represent changes relatively late in the disease process and leaves CAA in AD often undetected. Recently, it was shown that decreased vascular reactivity (VR) measured with blood oxygen level dependent (BOLD) MRI, after visual stimulus, is an early CAA marker. With BOLD-MRI to detect decreased VR in different stages of AD, it was shown that increasing stages of AD associate with decreasing VR independent of age, classic SVD markers and atrophy. Moreover, VR is associated with cognitive deficits. Therefore, cross-sectional data indicate that decreased VR is an important co-morbidity already in early stages of AD with an independent effect on disease severity. In this respect, the study aim is to determine the natural course of the decrease of VR in both controls and (early stage) AD patients to monitor AD disease progression. This is an essential step to aid in the development and application of effective treatment as it is expected that CAA can cause/worsen AD pathology.

DETAILED DESCRIPTION:
Rationale: Cerebral amyloid angiopathy (CAA), a common cerebrovascular small vessel disease (SVD), is a frequently (98%) found co-morbidity at autopsy in patients with Alzheimer's disease (AD). Current in vivo hallmarks of CAA represent changes relatively late in the disease process and leaves CAA in AD often undetected. Recently, it was shown that decreased vascular reactivity (VR) measured with blood oxygen level dependent (BOLD) MRI, after visual stimulus, is an early CAA marker. With BOLD-MRI to detect decreased VR in different stages of AD, it was shown that increasing stages of AD associate with decreasing VR independent of age, classic SVD markers and atrophy. Moreover, VR is associated with cognitive deficits. Therefore, cross-sectional data indicate that decreased VR is an important co-morbidity already in early stages of AD with an independent effect on disease severity. In this respect, the study aim is to determine the natural course of the decrease of VR in both controls and (early stage) AD patients to monitor AD disease progression. This is an essential step to aid in the development and application of effective treatment as it is expected that CAA can cause/worsen AD pathology.

Objective: To investigate longitudinal changes in VR in patients with subjective cognitive impairment (SCI), mild cognitive impairment (MCI) and AD dementia compared with controls. To investigate whether VR predicts progression of disease severity (cognitive decline) over a time period of 3 years and to investigate if decreased VR at baseline predicts increasing severity of other MRI markers for AD and SVD-markers at follow-up.

Study design: an longitudinal observational case - control study.

Study population: 30 AD patients, 30 patients with mild cognitive impairment and 30 patients with subjective cognitive impairment plus 30 controls, 50-90 yr old.

Main study parameters/endpoints: 1) 3T MRI: the amplitude of the BOLD response in percentage signal change between stimulus on and off, time-to-peak response (sec), and time-to-baseline (sec) after discontinuation of the visual stimulus, classic signs of CAA (intracranial hemorrhage, lobar microbleeds, subarachnoidal hemorrhage and superficial siderosis) and SVD markers (number of small subcortical infarcts and lacunes, volume of white matter hyperintensities (WMHs), perivascular spaces in the basal ganglia and centrum semiovale, number and location of deep microbleeds and grey matter volume). 2) Neuropsychological assessment 3) Baseline characteristics, 4) DNA: APOE ε genotype.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This is a non-therapeutic group relatedness study in only capacitated subjects. In order to achieve the aim of the study AD patients are needed. Vascular reactivity has potential to determine the role of the vascular aspects in AD. The risks of this research are minimal (risk of every day life), because there are no consequences to the health of the participant. We will keep the burden at a minimum. The research will consist of a 60 minutes MRI scan, a neuropsychological assessment of 1 hour and collection of 2 ml saliva (if not already collected at baseline).

ELIGIBILITY:
Inclusion Criteria:

* For this study three different routes for inclusion exists. Inclusion criteria for each group separately are shown below.

  1. Participants who were included in our previous CASCADE study (P19.039).

     * Capable of giving informed consent (see appendix)
  2. Patients who attended a memory clinic within one year ago

     * Diagnosed with (mixed) probable AD
     * Diagnosed as MCI
     * Diagnosed as SCI
     * Age between 50-90 years
     * Capable of giving informed consent (see appendix)
  3. Control subjects

     * Healthy adults without memory complaints
     * Age between 50 -90 years
     * Capable of giving informed consent

Exclusion Criteria:

* Contra-indication to MRI scanning:

  * Claustrophobia
  * Pacemakers and defibrillators
  * Nerve stimulators
  * Intracranial clips
  * Intraorbital or intraocular metallic fragments
  * Cochlear implants
  * Ferromagnetic implants
  * Hydrocephaluspump
  * Intra-utrine device (not all types) Permanent make-up
  * Tattoos above the shoulders (not all)
* Specific contraindications to fMRI

  * Seizure within prior year.
  * Noncorrectable visual impairment.
* MMSE < 19 points (measured at moment of screening or at memory clinic with a maximum of 6 months in retrospect)
* Severe physical restrictions (completely wheelchair dependent)
* Age above 90

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who attended a memory clinic and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Vascular reactivity - BOLD amplitude | 1,5 - 2 years between time point 1 and time point 2
  The change in BOLD signal in response to visual stimulation as measured by the amplitude of the BOLD response in percentage signal change between stimulus on and off.
Vascular reactivity - time-to-peak | 1,5 - 2 years between time point 1 and time point 2
  The time-to-peak response (sec) is defined as the duration from the beginning of visual stimulation to the peak response.
Vascular reactivity - time-to-baseline | 1,5 - 2 years between time point 1 and time point 2
  The time-to-baseline response (sec) is defined as the duration from the end of the stimulus to baseline.

SECONDARY OUTCOMES:
Intracranial hemorrhage | 1,5 - 2 years between time point 1 and time point 2
  number
Lobar microbleeds | 1,5 - 2 years between time point 1 and time point 2
  number
Subarachnoidal hemorrhage | 1,5 - 2 years between time point 1 and time point 2
  number
Superficial siderosis | 1,5 - 2 years between time point 1 and time point 2
  absent / focal / disseminated
Lacunes | 1,5 - 2 years between time point 1 and time point 2
  number
Volume of white matter hyperintensities (WMHs) | 1,5 - 2 years between time point 1 and time point 2
  cm3
Perivascular spaces in the basal ganglia | 1,5 - 2 years between time point 1 and time point 2
  degree 1: <5 PVS degree 2: 5 - 10 PVS degree 3: >10 PVS (but still numerable) degree 4: an innumerable number of PVS
Perivascular spaces in the centrum semiovale | 1,5 - 2 years between time point 1 and time point 2
  0= no PVS
  1. < 10 PVS
  2. 11-20 PVS
  3. 21-40 PVS
  4. >40 PVS
Gray matter volume | 1,5 - 2 years between time point 1 and time point 2
  cm3

CONTACTS AND LOCATIONS:
Locations (1):
- Leids Universitair Medisch Centrum, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided